CLINICAL TRIAL: NCT03572946
Title: Diagnostic Efficiency With Magnetic Resonance Imaging-targeted Biopsy Compared to Standard Transperineal Ultrasound-guided Biopsy in Biopsy-naïve Suspicious Prostate Cancer Patients: A Randomized Controlled Trial
Brief Title: Targeted Biopsy or Standard Biopsy for Clinical Significant Prostate Cancer Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Biopsy Protocol v2.0 20181009
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2018-10

CONDITIONS: Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- target biopsy group (Experimental): Targeted prostate biopsy
  Interventions: Procedure: Targeted prostate biopsy
- standard biopsy group (Active Comparator): Standard prostate biopsy
  Interventions: Procedure: Standard biopsy

INTERVENTIONS:
Procedure: Targeted prostate biopsy — MRI-guided targeted prostate biopsy
  Arms: target biopsy group
Procedure: Standard biopsy — Transperineal ultrasound guided prostate biopsy(SB).
  Arms: standard biopsy group

SUMMARY:
This randomized controlled trial aims to assess the detection rate of clinically significant and clinically insignificant cancer of mpMRI-targeted biopsy compared to transperineal standard biopsy in men with clinical suspicion of prostate cancer who had no prior prostate biopsy.

DETAILED DESCRIPTION:
Prostate biopsy with multiple samples using a standardized template (standard biopsy, SB) under transrectal ultrasound (TRUS) guidance is the current standard diagnostic approach in suspicion of prostate cancer (PCa). However, many biopsies are unnecessary or cannot detect clinically significant PCa (csPCa).

With the introduction of multiparametric magnetic resonance imaging (mpMRI) of the prostate and the improvement for PCa detection and localization, an alternative procedure, known as MRI-targeted biopsy (TB), has been shown comparable or even higher detection rates of csPCa compared to TRUS-biopsy (SB).

This randomized controlled trial aims to assess the detection rate of clinically significant and clinically insignificant cancer of TB compared to SB (transperineal) in men referred with clinical suspicion of prostate cancer who have had no prior prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Men more than 18 years old with clinical suspicion of prostate cancer;
2. Serum PSA ≤ 20 ng/ml within the previous 3 months;
3. Suspected stage ≤ T2 on rectal examination (organ-confined prostate cancer) within the previous 3 months;
4. No evidence of PSA increase by noncancerous factors, such as catheterization, bladder stones, or urinary tract infection including bacterial prostatitis;
5. mpMRI PI-RADS V2 score 4 or 5；
6. Able to provide written informed consent.

Exclusion Criteria:

1. Prior prostate biopsy or prostate surgery;
2. Prior treatment for prostate cancer;
3. Contraindication to MRI (e.g. claustrophobia, pacemaker, estimated glomerular filtration rate ≤ 50mls/min);
4. Contraindication to prostate biopsy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Detection rates of clinically significant PCa | 30 days post biopsy
  Clinically significant prostate cancer is considered as: biopsy Gleason score ≥3+4 or maximum cancer core length ≥5 mm.

SECONDARY OUTCOMES:
Detection rates of clinically insignificant PCa | 30 days post biopsy
  Clinically insignificant prostate cancer is considered as: biopsy Gleason score <3+4 and maximum cancer core length <5 mm.
Biopsy-related adverse events | 30 days post biopsy
Proportion of men undergoing radical prostatectomy who have Gleason grade upgrading | 90 days post-biopsy
  Comparing the Gleason grades (from 1-5, the bigger the worse) between biopsy and final pathology, Gleason grade is upgrading when the Gleason grade of final pathology is bigger than that of biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, PhD, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China